CLINICAL TRIAL: NCT01873573
Title: Randomized Controlled Trial of Endoscopic Dilation With or Without Triamcinolone Injection in Patients With Non-malignant Radiation or Anastomotic Esophageal Strictures
Brief Title: Randomized Controlled Trial of Endoscopic Dilation: Triamcinolone Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17316
Record Dates: First submitted 2013-06-04; First posted 2013-06-10 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Dysphagia
Keywords: radiation-induced stricture; anastomotic stricture; esophagogastroduodenoscopy (EGD); dilation; steroid injection; triamcinolone; difficulty swallowing
MeSH Terms: conditions — Deglutition Disorders; Dilatation, Pathologic | interventions — Dilatation; Triamcinolone; Steroids; Adrenal Cortex Hormones; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGD with Dilation (Active Comparator): Standard of Care: Esophagogastroduodenoscopy (EGD) with dilation alone. If participants are assigned to Arm A and are not showing any clinical improvements as determined by their physician after the first three endoscopic dilation sessions, then they will be crossed over into Arm B.
  Interventions: Procedure: Dilation; Procedure: Esophagogastroduodenoscopy (EGD)
- EGD with Dilation, plus Triamcinolone (Active Comparator): Standard of Care: EGD with dilation and Triamcinolone injection.
  Interventions: Procedure: Dilation; Other: Triamcinolone Injection; Procedure: Esophagogastroduodenoscopy (EGD)

INTERVENTIONS:
Procedure: Dilation — Dilation will be performed by either dilation balloons or over the wire polyvinyl dilators based upon the physician's discretion. Fluoroscopy may be used to aid in endoscopic dilation at the physician's discretion.
Other: Triamcinolone Injection — Triamcinolone is a generic name of a long-acting synthetic corticosteroid and approved for sale in the United States by the U.S. Food and Drug Administration (FDA). After endoscopic dilation is performed, a total of 40-80 mg (physician preference) of triamcinolone (40 mg/ml) will be injected throughout the stricture under direct visualization.
  Other Names: steroid; corticosteroid; Kenalog 10
  Arms: EGD with Dilation, plus Triamcinolone
Procedure: Esophagogastroduodenoscopy (EGD) — EGD is a test to examine the lining of the esophagus (the tube that connects your throat to your stomach), stomach, and first part of the small intestine. It is done with a small camera (flexible endoscope) that is inserted down the throat.
  Other Names: flexible endoscope

SUMMARY:
The purpose of this pilot study is to find out if adding triamcinolone (steroid) injection at the participant's initial esophagogastroduodenoscopy (EGD) procedure will improve the opening of their esophagus and decrease the need for repeat dilations.

DETAILED DESCRIPTION:
This is a randomized two-arms cross-over trial. In this study there are two groups, the control group and the triamcinolone treatment group. The cross-over design will apply only in the control group when patients are not responding to EGD dilations alone (defined as no sustained improvement in baseline dysphagia) and they will be allowed to cross-over to the triamcinolone group and undergo 3 successive EGDs with triamcinolone injection.

Typically, triamcinolone (steroid) injection is given as a standard of care after several esophageal dilations are performed and failed to improve the condition. Therefore, researchers want to find out if adding triamcinolone (steroid) injection at the participant's initial EGD procedure will improve the opening of their esophagus and decrease the need for repeat dilations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present for EGD with dilation for dysphagia symptoms thought secondary to either radiation-induced stricture or anastomotic stricture based on history

Exclusion Criteria:

* Inability to consent for the procedure
* Known coagulopathy [International Normalized Ratio (INR) >1.5, Platelets <75 K]
* Endoscopic finding of a stricture that is not caused by either radiation or anastomotic narrowing
* Nasopharyngeal strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Number of Visits to Receive Esophageal Dilation During the 12 Month Follow-up Period | 12 months
  The main outcome measured will be number of visits to receive Esophageal Dilation during the 12-month follow-up period. Successful dilation of the stricture for the procedure will be defined as creation of a mucosal tear confirmed by endoscopic visualization after the last dilation is performed.

SECONDARY OUTCOMES:
Final Dysphagia Score | 12 months
  Dysphagia Scoring System: 0 = able to eat normal diet / no dysphagia; 1 = able to swallow some solid foods; 2 = able to swallow only semi solid foods; 3 = able to swallow liquids only; 4 = unable to swallow anything / total dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Klapman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States